CLINICAL TRIAL: NCT04784910
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DWP14012 in Prevention of NSAIDs Induced Peptic Ulcer
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 in Prevention of NSAIDs Induced Peptic Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DW_DWP14012304
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — fexuprazan; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP14012 20mg (Experimental): orally, once daily
  Interventions: Drug: DWP14012 20mg; Drug: Lansoprazole 15 mg placebo
- Lansoprazole 15mg (Active Comparator): orally, once daily
  Interventions: Drug: Lansoprazole 15 mg; Drug: DWP14012 20mg placebo

INTERVENTIONS:
Drug: DWP14012 20mg — DWP14012 20mg, tablet, orally, once daily for up to 24 weeks
  Arms: DWP14012 20mg
Drug: Lansoprazole 15 mg — Lansoprazole 15mg capsule, orally, once daily for up to 24 weeks
  Arms: Lansoprazole 15mg
Drug: DWP14012 20mg placebo — DWP14012 20mg placebo-matching tablet, orally, once daily for up to 24 weeks
  Arms: Lansoprazole 15mg
Drug: Lansoprazole 15 mg placebo — Lansoprazole 15mg placebo matching capsule, orally, once daily for up to 24 weeks
  Arms: DWP14012 20mg

SUMMARY:
The study aims to demonstrate the preventive effect of DWP14012 20 mg for peptic ulcer is non-inferior to that of Lansoprazole 15 mg in terms of prevention of peptic ulcer and confirm the safety of DWP14012 20 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged ≥ 19 years at the time of informed consent
2. Subjects who are diagnosed with musculoskeletal disease at screening and require continued treatment with NSAIDs for at least 24 weeks
3. Subjects with at least one of the following risk factors for ulcer development at screening.
4. Subjects who have no gastric or duodenal mucosal break or have ulcer in the scarring stage based on the EGD result at screening.

Exclusion Criteria:

1. Subjects with esophagitis, gastroesophageal varix, esophagus, Barrett's esophagus, acute gastrointestinal bleeding and else based on the screening EGD results.
2. Subjects who have undergone gastroduodenal surgery or total small bowel resection
3. Subjects with history of clinically significant disease of hepatic, renal, nervous, pulmonary, endocrine, hemato-oncologic, cardiovascular or urinary system
4. Subjects who have had a malignant tumor in the last 5 years
5. Subjects who history of hypersensitivity to the IP ingredients, aspirin and NSAIDs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who develop peptic ulcer by Week 24 as assessed by investigator | at 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects who develop peptic ulcer by Week 12 as assessed by investigator | at 12 weeks
Proportion of subjects with endoscopic gastric or duodenal bleeding** by Week 12 and Week 24 | at 12, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong S, Ju JH, Lee SH, Hong SJ, Kim SH, Ahn GY, Jung JH, Hur JW, Ha YJ, Park JK, Kim HS, Lee SW, Park YB, Lim MJ, Kim YS, Song JS, Choi CB, Kim SH, Choi IA, Choi KD, Lee TH, Cho YS, Lee YC, Kwon KS, Lee H, Park M, Heo J, Baek S, Lee CK. Comparing the Efficacy and Safety of Fexuprazan and Lansoprazole for the Prevention of Nonsteroidal Anti-inflammatory Drug-Induced Peptic Ulcer. Gut Liver. 2025 Sep 15;19(5):685-695. doi: 10.5009/gnl250019. Epub 2025 Jun 26. PMID 40567214